CLINICAL TRIAL: NCT04697563
Title: Laser Therapy in Women With Lichenoid Disorders: A Randomized Controlled Trial
Brief Title: Laser Therapy in Women With Lichenoid Disorders
Acronym: Liser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Liser
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Lichen Sclerosus Et Atrophicus; Lichen Planus
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus; Lichen Planus | interventions — Lasers

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded placebo- controlled clinical study
Who Masked: Participant, Investigator
Masking Description: The person who performs the laser treatment is unaware of the treatment given The laser devices can be used as a placebo laser by blocking the laser beam with a plug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laser (Active Comparator): Before treatment the vulva will be carefully inspected to rule out signs of infection or recent trauma. A local anesthetic cream (Emla cream 5%) will be applied to the entire introitus vulvae and all areas intended for local laser treatment. Before laser treatment another cotton swab test will be performed to ensure sufficient local anesthesia.
  Vulvovaginal laser therapies will be performed with the non-ablative 2940 nm Er:YAG laser (Smooth XS, Fotona, Slovenia) in the Renova mode according to the manufacturer's guidelines and recommendations. The spot size (diameter of the laser beam) is 7 mm, with a pulse at a frequency of 1.6 Hz, and a fluence (laser energy delivered per unit area) of 5.0 to 10.0 J/cm2. The vulva will be treated using 1-3 repetitions.
  Interventions: Device: Laser
- Placebo Laser (Placebo Comparator): Clinical examination and preparations will be identical to the intervention group. Sham laser treatments will be performed with the same laser and the same device. However, a specially designed placebo probe, which blocks the emission of radiation, will be used. Women will therefore receive no therapeutic laser treatment. Before treatment, a study assistant, who is aware of the study allocation, will prepare the laser with the placebo probe, which looks identically to the "normal" probe. The treating physician will not be aware of the study allocation and the type of probe in use.
  Interventions: Device: Placebolaser

INTERVENTIONS:
Device: Laser — real laser beam administered
  Other Names: Fotona Smooth XS laser
  Arms: Laser
Device: Placebolaser — no laser beam admitted
  Other Names: Fotona Smooth XS laser placebo
  Arms: Placebo Laser

SUMMARY:
Primary aim of the trial is to compare improvement of lichen symptoms according to a composite VAS scale (burning, itching and pain) between women with vulvovaginal laser therapy vs. sham laser therapy at three months.

DETAILED DESCRIPTION:
Background: Lichenoid Disorders (LD) include VLS (Vulvar lichen sclerosus) and LP (Lichen planus). VLS and LP are chronic skin diseases that usually affect the anogenital region. Both can cause vulvar itching, burning and pain and can lead to urinary and sexual dysfunction. Current treatment options are unsatisfactory. Vulvovaginal laser therapy might be an effective treatment option.

Study aim: To study the effectiveness of non-ablative vulvovaginal laser therapy for women with lichenoid disorders.

Design: Randomized double-blinded placebo- controlled clinical study

Study Population: Women diagnosed with LD will be recruited from a specialized University outpatient clinic.

Study groups: Participants will be randomized (1:1). Intervention group: Laser therapy (2 treatments), plus ongoing therapy Control group: Sham laser therapy (2 treatments) plus ongoing therapy

Sample size Total 40 patients Primary study outcome: Visual analogue scale (VAS) composite score in regard to LD Secondary study outcomes: quality of life (QoL) (Skindex questionnaire); Treatment discomfort/ pain (VAS); Patient treatment satisfaction (Questionnaire to ask for treatment satifsaction: ZUF-8); Subjective improvement (Patient global impression of improvement- PGI-I), clinical LS score, histological appearance

ELIGIBILITY:
Inclusion criteria

* women age >18 years
* diagnosed with LD (VLS or LP histologically proven)
* Clinical LS score ≥ 4 based on the score of Günthert et al. [1]
* Normal Pap-smear within 24 months
* negative clinical and microscopic evaluation of vaginal fluid
* Negative test for STD (sexually transmitted diseases) pathogens (chlamydia, gonorrhea, genital mycoplasma and trichomonas) if symptomic including abdominal pain or abnormal vaginal fluid
* Good German language skills
* written informed consent
* preceding local corticoid therapy of at least 12 weeks according to the current guideline for LD

Exclusion criteria:

* women with contraindications for the use of laser on the skin
* pregnancy
* presence of vulvar pathology (other than lichen)
* any vulvar/ vaginal infection
* immunocompromised women
* swollen lymph nodes
* genital malignant disease
* allergy to topical anaesthesia
* connective tissue disease
* keloid formation
* Patients with a legal guardian
* Body Mass Index > 35 kg/m²
* History of transvaginal mesh implant (excluding sling or sacrocolpopexy mesh)
* Coagulopathy
* patients using anticoagulants
* patients with renal, hepatic or pulmonary-cardiovascular failure
* patients who have undergone any kind of organ transplantation in the last three years.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — only females can participate in this study because it is lead by gynecologists
Enrollment: 40 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
subjective bother of lichenoid disorders (LD) | 3 months
  A visual analogue scale (VAS) is used for assessment for the subjective bother of LD symptoms. Patients are asked to indicate the degree of each of the three following LD symptoms on a scale ranging from 0 (no symptoms) to 10 (worst possible symptoms):
  genital symptoms of itching, burning and vaginal pain resulting in a composite VAS score

SECONDARY OUTCOMES:
Treatment discomfort / pain | 3 months
  patients are asked to indicate the degree of discomfort or pain during laser therapy on a visual analogue scale (VAS) ranging from 0 (no discomfort/pain) to 10 (worst possible discomfort/pain)
subjective symptoms of lichenoid disorders | 3 months
  The Skindex questionnaire will be used to evaluate patients' subjective symptoms of lichenoid disorders
Patient Global Impression of Improvement- PGI-I | 3 months
  The PGI-I scales are robust and valid instruments to assess disease severity, bother and improvement after treatment in women and will be used to determine the Patient Global Impression of Improvement. The PGI-I consists of a 7-likert-scale with 7 being the worst bother.
Patient Global Impression of Severity- PGI-S | 3 months
  The Patient Global Impression of Severity (PGI-S) is a global index that may be used to rate the severity of a specific condition (a single-state scale). The PGI scales are robust and valid instruments to assess disease severity, bother and improvement after treatment and will be used to determine the Patient Global Impression of Severity. The PGI scales are robust and valid instruments to assess disease severity, bother and improvement after treatment. The patient can choose from 4 answers including none, mild, moderate and severe.
architectural changes | 3 months
  The vulva will be inspected and structural changes due to LD will be recorded. The score is based on the publication from Günthert et al. The score records signs of erosions, hyperkeratosis, rhagades, synechia, stenosis, and atrophy of the vulva. The questionnaires is based on a 29-item version; the higher the score the more pronounced are the clinical signs.
Histological analysis of LD | 3 months
  Lichenoid disorders show epidermic atrophy, sclerosis and a lymphocytic based dermal inflammation. Hyperkeratosis and dermal inflammation will be evaluated both from the histological probe before and after treatment. Each item will be scored from 1-3, mild, moderate and severe. A higher score indicates more severe expression of LD.
Patient satisfaction with treatment/ inpatient management | 3 months
  Patient satisfaction will be evaluated with the "Fragebogen zur Patientenzufriedenheit - ZUF8". The German version of the original "Client Satisfaction Questionnaire-CSQ8", is a validated tool for measuring global patient satisfaction at the end of inpatient treatment. he Zuf-8 is an 8-items questionnaire to assess satisfaction in patients undergoing inpatient treatment. At 3 months treatment satisfaction will be assessed using an adopted version of the questionnaire. The lower the score the higher is the patient satiscation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics, Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No